CLINICAL TRIAL: NCT04561531
Title: Efficacy and Safety of Intermittent Bolus Comparing With Traditional Continuous Drip of 3% NaCl in Patients With Severe Symptomatic Hyponatremia at Rajavithi Hospital
Brief Title: Efficacy and Safety of Bolus Comparing With Continuous Drip of 3% NaCl in Patients With Severe Symptomatic Hyponatremia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 148/2563
Record Dates: First submitted 2020-08-28; First posted 2020-09-23 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-08

CONDITIONS: Hyponatremia; Osmotic Demyelination Syndrome
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent bolus (Experimental): In intermittent bolus of 3%NaCl group ,patients will receive intermittent bolus of 3%NaCl 150 ml in 30 minutes and then follow plasma sodium,observe glasglow coma scale and level of consciousness until improvement of consciousness and achieve target plasma sodium which is 5 mmol/L in 6 hours and should not be overcorrected which defined that plasma sodium change should not be more than 12 mmol/L in 24 hours and 18 mmol/L in 48 hours.
  Interventions: Other: 3%NaCl
- Traditional continuous drip (Experimental): In traditional continuous drip of 3%NaCl group ,patients will receive 3%NaCl adjust rate start from 1 ml/kg/hr and follow plasma sodium every 1 hour,observe glasglow coma scale and level of consciousness until improvement of consciousness and achieve target plasma sodium which is 5 mmol/L in 6 hours and should not be overcorrected which defined that plasma sodium change should not be more than 12 mmol/L in 24 hours and 18 mmol/L in 48 hours.
  Interventions: Other: 3%NaCl

INTERVENTIONS:
Other: 3%NaCl — Intervention is infusion of 3%NaCl which is defined in arms of experiment.

SUMMARY:
To compare between intermittent bolus and traditional continuous drip of 3%NaCl in patients with severe symptomatic hyponatremia in Rajavithi Hospital.

DETAILED DESCRIPTION:
Background: Hyponatremia is the most common electrolyte imbalance in clinical practice, associated with increased mortality and length of stay. In 2014,European guideline have recommended promp infusion of 3%NaCl 150 ml in 20 minutes to raise plasma Na to 5 mmol/L and improve symptoms. The recommendation was the result of studies with small numbers of patients, and expert opinions.

Methods: A single center opened-label randomized controlled-trial,we will randomly assign 40 patients with severe symptomatic hyponatremia (plasmaNa<125mmol/L) in Rajavithi Hospital into two groups:

First group receive intermittent bolus of 3%NaCl 150 ml in 30 minutes and follow plasma sodium until achieve target of goal plasma sodium = 5 mmol/L in 6 hours (no more than 12 mmol/L in 24 hr and 18 mmol/L in 48 hr),another receive traditional continuous drip of 3%NaCl start with rate = 1ml/kg/hr and follow plasma sodium every 1 hour until achieve target of plasma sodium 5 mmol/L in 6 hours .The primary end point is change in plasma sodium in 6 hours and improvement of glasglow coma scale.The secondary end points are change in plasma sodium in 24,48 hours,overcorrection rate in 24 and 48 hours ,ODS rate ,hospitality days and mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Rajavithi Hospital
* Age from 18 years
* Plasma Na < 125 mmol/l with glucose-corrected
* Severe symptomatic hyponatremia (Vomitting ,Coma ,Somnolence)

Exclusion Criteria:

* Systolic BP < 90 mmHg Or MAP< 70 mmHg
* Pregnancy or Lactation
* Congestive Heart Failure or Volume overload
* Lung congestionfrom CXR
* Chronic renal failure patients with edema
* Cirrhosis patients with edema
* Patients with coronary artery disease
* Patients with brain injuries
* Deny consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Plasma sodium and glasglow coma scale(GCS) | 6 hours
  Change in plasma sodium and level of consciousness (GCS)

SECONDARY OUTCOMES:
Plasma sodium and glasglow coma scale(GCS) | 24 and 48 hours
  Change in plasma sodium and level of consciousness (GCS)
overcorrection rate | 24 and 48 hours
  rate of overcorrection which defined as change in plasma sodium over 12 mmol/L in 24 hr and 18 mmol/L in 48 hr
ODS rate | in 7 days
  rate of osmotic demyelinating syndrome
hospitality days | until discharge
  hospitality days
mortality rate | in 30 days
  mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King JD, Rosner MH. Osmotic demyelination syndrome. Am J Med Sci. 2010 Jun;339(6):561-7. doi: 10.1097/MAJ.0b013e3181d3cd78. PMID 20453633
- [Result] Spasovski G, Vanholder R, Allolio B, Annane D, Ball S, Bichet D, Decaux G, Fenske W, Hoorn EJ, Ichai C, Joannidis M, Soupart A, Zietse R, Haller M, van der Veer S, Van Biesen W, Nagler E; Hyponatraemia Guideline Development Group. Clinical practice guideline on diagnosis and treatment of hyponatraemia. Eur J Endocrinol. 2014 Feb 25;170(3):G1-47. doi: 10.1530/EJE-13-1020. Print 2014 Mar. PMID 24569125
- [Result] Ayus JC, Krothapalli RK, Arieff AI. Treatment of symptomatic hyponatremia and its relation to brain damage. A prospective study. N Engl J Med. 1987 Nov 5;317(19):1190-5. doi: 10.1056/NEJM198711053171905. PMID 3309659
- [Result] Adrogue HJ, Madias NE. Hyponatremia. N Engl J Med. 2000 May 25;342(21):1581-9. doi: 10.1056/NEJM200005253422107. No abstract available. PMID 10824078
- [Result] Ball SG, Iqbal Z. Diagnosis and treatment of hyponatraemia. Best Pract Res Clin Endocrinol Metab. 2016 Mar;30(2):161-73. doi: 10.1016/j.beem.2015.12.001. Epub 2015 Dec 30. PMID 27156756
- [Result] Sterns RH, Nigwekar SU, Hix JK. The treatment of hyponatremia. Semin Nephrol. 2009 May;29(3):282-99. doi: 10.1016/j.semnephrol.2009.03.002. PMID 19523575
- [Result] Koenig MA, Bryan M, Lewin JL 3rd, Mirski MA, Geocadin RG, Stevens RD. Reversal of transtentorial herniation with hypertonic saline. Neurology. 2008 Mar 25;70(13):1023-9. doi: 10.1212/01.wnl.0000304042.05557.60. Epub 2008 Feb 13. PMID 18272864
- [Result] Hoorn EJ, Zietse R. Diagnosis and Treatment of Hyponatremia: Compilation of the Guidelines. J Am Soc Nephrol. 2017 May;28(5):1340-1349. doi: 10.1681/ASN.2016101139. Epub 2017 Feb 7. PMID 28174217
- [Result] Garrahy A, Dineen R, Hannon AM, Cuesta M, Tormey W, Sherlock M, Thompson CJ. Continuous Versus Bolus Infusion of Hypertonic Saline in the Treatment of Symptomatic Hyponatremia Caused by SIAD. J Clin Endocrinol Metab. 2019 Sep 1;104(9):3595-3602. doi: 10.1210/jc.2019-00044. PMID 30882872
- [Result] George JC, Zafar W, Bucaloiu ID, Chang AR. Risk Factors and Outcomes of Rapid Correction of Severe Hyponatremia. Clin J Am Soc Nephrol. 2018 Jul 6;13(7):984-992. doi: 10.2215/CJN.13061117. Epub 2018 Jun 5. PMID 29871886
- [Result] Mohmand HK, Issa D, Ahmad Z, Cappuccio JD, Kouides RW, Sterns RH. Hypertonic saline for hyponatremia: risk of inadvertent overcorrection. Clin J Am Soc Nephrol. 2007 Nov;2(6):1110-7. doi: 10.2215/CJN.00910207. Epub 2007 Oct 3. PMID 17913972
- [Result] Owen BE, Rogers IR, Hoffman MD, Stuempfle KJ, Lewis D, Fogard K, Verbalis JG, Hew-Butler T. Efficacy of oral versus intravenous hypertonic saline in runners with hyponatremia. J Sci Med Sport. 2014 Sep;17(5):457-62. doi: 10.1016/j.jsams.2013.09.001. Epub 2013 Sep 18. PMID 24148616
- [Result] Lee A, Jo YH, Kim K, Ahn S, Oh YK, Lee H, Shin J, Chin HJ, Na KY, Lee JB, Baek SH, Kim S. Efficacy and safety of rapid intermittent correction compared with slow continuous correction with hypertonic saline in patients with moderately severe or severe symptomatic hyponatremia: study protocol for a randomized controlled trial (SALSA trial). Trials. 2017 Mar 29;18(1):147. doi: 10.1186/s13063-017-1865-z. PMID 28356136
- See also: 7. Mohamed OH, Abdallah N. Prevention and treatment of the osmotic demyelination syndrome: JSM Brain Sci 2016; 1: 1004. — http://www.jscimedcentral.com/BrainScience/brainscience-1-1004.pdf
- See also: 14. Lambeck J, Hieber M, Dreßing A, Niesen WD. Central pontine myelinolysis and osmotic demyelination syndrome. Dtsch Arztebl Int. 2019; 116: 600-6. — https://www.aerzteblatt.de/int/archive/article/209401/Central-pontine-myelinolysis-and-osmotic-demyelination-syndrome